CLINICAL TRIAL: NCT05430776
Title: The Effect of Systemic Versus Local Transcutaneous Laser Therapy on Tension-type Cephalea and Orofacial Pain in Post-covid-19 Patients: a Pragmatic Randomized Clinical Trial.
Brief Title: Laser Therapy on Tension-type Cephalea and Orofacial Pain in Post-covid-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Lara Jansiski Motta, PhD, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBMPOSTCOVID
Record Dates: First submitted 2022-06-22; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Tension-Type Headache; Orofacial Pain; COVID-19
Keywords: tension-type headache; orofacial pain; photobiomodulation; covid-19
MeSH Terms: conditions — Tension-Type Headache; Facial Pain; COVID-19

STUDY DESIGN:
Intervention Model Description: 2 groups systemic versus local transcutaneous laser therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local photobiomodulation (Active Comparator): photobiomodulation with red and infrared laser with local application on pain points and
  Interventions: Radiation: Photobimodulation
- Systemic photobiomodulation (Experimental): photobiomodulation with red laser with transcutaneous application in the radial artery.
  Interventions: Radiation: Photobimodulation

INTERVENTIONS:
Radiation: Photobimodulation — laser therapy application

SUMMARY:
Considering the auxiliary potential effect of photobiomodulation in controlling persistent CTT and TMD-related pain in patients who have been diagnosed with COVID-19, and are recovered from the viral infection, we intend to conduct a clinical trial comparing two modalities of therapeutic laser application: local application and transcutaneous application in the radial artery.

One of the main advantages of auxiliary techniques in pain control is the decrease of the use of drugs for analgesia, avoiding side effects and tolerance caused by them, and promoting an improvement in the individual's quality of life.

DETAILED DESCRIPTION:
Orofacial pain and tensional cephalea were symptoms commonly reported in COVID-19 patients, even after recovery, and were considered chronic pain in these cases. The pain control, in these cases, is mostly accomplished with the use of analgesic and anti-inflammatory drugs. However, there are auxiliary treatments that can reduce the amount of pharmacological intake and improve the quality of life of compromised individuals, one of them is photobiomodulation. Using lasers for treatments to control inflammation and pain is successfully performed, but the parameters and the ways of application are not yet strongly established. The aim of this research is to evaluate the effect of the application of photobiomodulation with red and infrared lasers applied locally and systemically. For this purpose, individuals who have been diagnosed with COVID-19 and have had a tension headache and/or orofacial pain for more than 3 months will be selected by convenience. The participants will be divided into two different groups: G1- photobiomodulation with red and infrared laser with local application on the pain points (808 nm and 660 nm,100 mW, 6J per point) and G2 -photobiomodulation with red laser with transcutaneous application on the radial artery (660 nm, 100mW, 30 minutes). All participants will be treated for a period of 4 weeks, with 8 application sessions. The effects will be measured by means of blood lactate level, Brief Pain Inventory, Visual Analog Scale (VAS), and Cephalea Impact Test.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes, between the ages of 19 and 65, complaining of persistent orofacial pain or functional-type cephalea, for more than 3 months.
* Individuals diagnosed with COVID-19, confirmed by RT-PCR for SARS-CoV-2 already recovered, at least 30 days after infection.

Exclusion Criteria:

* Individuals with diagnoses of neuropathies and headaches other than tension-type headache
* Physical or intellectual incapacity to answer the survey questionnaires; illiterate; diabetics, pacemakers, and pregnant women.
* Individuals who report photosensitivity to laser.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
headache and orofacial pain | four weeks
  headache and orofacial pain by analogic visual escale

CONTACTS AND LOCATIONS:
Overall Officials: Lara Motta, Phd, Principal Investigator — Nove de Julho University
Locations (2):
- Brazil (2):
  - Nove de Julho Univ, São Paulo, São Paulo
  - Lara Motta, São Roque, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costanti Vilela Campos M, Simoes Velloso Schuler S, de Barros Motta P, Catia Mazzoni A, Cristina da Silva F, Domingues Martins M, Porta Santos Fernandes K, Agnelli Mesquita-Ferrari R, Ratto Tempestini Horliana AC, Kalil Bussadori S, Jansiski Motta L. The effect of systemic versus local transcutaneous laser therapy on tension-type cephalea and orofacial pain in post-COVID-19 patients: A pragmatic randomized clinical trial. Medicine (Baltimore). 2022 Nov 18;101(46):e31218. doi: 10.1097/MD.0000000000031218. PMID 36401476